CLINICAL TRIAL: NCT00568971
Title: Phase II Study of Weekly Docetaxol Combined With Cisplatin and 5-Fu in Patients With Advanced Gastric Cancer
Brief Title: Study of Weekly DCF to Treat Advanced Gastric Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has finished.
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University cancer hospital, Fudan University cancer hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCF-AGC
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2009-08

CONDITIONS: Gastric Cancer
Keywords: DCF; Advanced gastric cancer; Phase II study; Efficacy; Toxicity
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- weekly chemo (Experimental): Docetaxel 33.3 mg/m2, Cisplatin 30 mg/m2 and 5-FU 1500 mg/m2 of 24-hour continuous intravenous infusion;d1,8,15 q4w.The treatment will not stopped until disease progression or unaccepted toxicities.
  Interventions: Drug: Docetaxel, Cisplatin, 5-Fu

INTERVENTIONS:
Drug: Docetaxel, Cisplatin, 5-Fu — Docetaxel 33.3 mg/m2, Cisplatin 30 mg/m2 and 5-FU 1500 mg/m2 of 24-hour continuous intravenous infusion;d1,8,15 q4w.The treatment will not stopped until disease progression or unaccepted toxicities.
  Other Names: wDCF

SUMMARY:
The purpose of this study is to evaluate the efficacy of weekly docetaxol combined with cisplatin and 5-Fu in patients with AGC.

DETAILED DESCRIPTION:
Recently,in a multi-center, open-label randomized phase III study (V325), compared to the control arm of CF regimen, DCF showed higher efficacy in terms of response rate, time to progression and overall survival. But the regimen had increased grade 3-4 neutropenia (82% vs 57%) and febrile neutropenia infection (29% vs 12%). We began to study on weekly DCF in the patients with advanced gastric cancer to evaluate the efficacy no less than that of 3-week' regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Patients with histologically confirmed, unresectable, recurrent and/or metastatic gastric adenocarcinoma
* ECOG performance status ≤1,life expectancy more than 3 months,
* Normal laboratory findings:absolute neutrophil count and platelet count ≥ 2.0×109/L and 80×109/L, respectively, hepatic function (total serum bilirubin ≤ UNL, transaminases ≤ 1.5 times upper normal limit) and renal function (calculated creatinine clearance ≥ 60 ml/min).
* Measurable disease according to the RECIST.

Exclusion Criteria:

* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection
* The evidence of CNS metastasis
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Received other chemotherapy regimen after metastasis
* Used taxane in adjuvant settings
* Participated in other clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Response rate, overall survival | 2-6 months

SECONDARY OUTCOMES:
Side effects | 2-6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China